CLINICAL TRIAL: NCT01441908
Title: Determining Cardiovascular Health Using a Multi-Analyte Profile in a Longitudinal Study of a Statin Intervention for Dyslipidemia
Brief Title: Longitudinal Study of Multi-Analyte Profile for Dyslipidemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MaiHealth Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MAI-001; 6R44HL082382-0 (Other Grant/Funding Number: SBIR); 6R44HL082382 (NIH)
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Dyslipidemia
Keywords: Cardiovascular; Multi-analyte; Statin; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control Group
- Statin (Active Comparator): Receiving Statin
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — 40mg or 80mg dose 28 days for 6 month period
  Arms: Statin

SUMMARY:
The primary objective of this study is to determine any changes in cardiovascular risk among individuals receiving a statin by assessing their multi-analyte profile.

DETAILED DESCRIPTION:
Over the past decade there has been a growing debate about the clinical value content of a single individual diagnostic indicator of disease onset, progression or therapeutic intervention. In particular there has been a discussion about the comparative value of a single biomarker versus a panel (3-6 different analytes) versus a multi-analyte profile (>10 different analytes) of biomarkers to provide high content clinical information about a specific disease onset, progression, remediation or treatment efficacy.

With the advent of personalized medicine, and recognition of the high degree of biological variability in human pathobiology, it is important to understand the comparative value of a single biomarker/diagnostic versus a panel versus a profile. In addition, the growth of Preventive Medicine has spurred the development of "Wellness" in individual patients, and the necessity for understanding and measuring the transition from a state of health (wellness) to ultimately a state of full blown disease onset. This complex process occurs via a multitude of biological pathways and networks and manifests at a biochemical and clinical systems level.

In a previous study currently being analyzed, MaiHealth measured a Multi-Analyte Profile of approximately 800 patients consisting of 400 cardiovascular compromised individuals and 400 control patients. This preliminary study was a single time point only, in which 25 individual analytes were measured as well as 3 calculated ratios or values for the 800 individuals.

The current study is a small cohort time course study over 6 months involving therapeutic intervention with an FDA-approved statin.

The overall goal of the study is to determine the predictive capability of a single versus panel versus multi-analyte profile set of biomarkers in cardiovascular compromised patients with therapeutic intervention. The ultimate application of this research is information delivery and behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sign and Date IRB approved consent form
* Be between 30-65 years of age as of date of consent
* Have a total cholesterol value of 200-300 (units)
* Have an LDL cholesterol value of > 100 (units)
* Able to speak and understand English
* Willing and able to participate for the 6 months required by the study
* Willing and able to provide fasting blood specimens
* Women of child-bearing potential must have a negative pregnancy test at screening
* Medically (appropriate) eligible to take the statin as determined by PI

Exclusion Criteria:

* Have a body Mass Index (BMI) > or = 35
* Pregnant (or planning to become pregnant during the course of the study)
* Currently taking a statin or discontinued taking a statin within 9 months of the date of screening

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of 29 specific cardiovascular related lab assays from baseline through a period of 6 months in a control population with dyslipidemia vs a study group with dyslipidemia receiving an FDA approved Statin (Pravastatin). | 6-month
  Comparative, predictive capability of a single versus panel versus multi-analyte profile for improvement in cardiovascular health as a function of therapeutic intervention over time. Comparative analyses will be performed against the control profile to track blood chemistry changes as a result of intervention.

SECONDARY OUTCOMES:
Limited time-course of different stages of disease regression | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Harper, MD, Principal Investigator — Wake Research Associates; Stephen Naylor, Ph.D., Study Director — MaiHealth Inc
Locations (1):
- Wake Research Associates, Raleigh, North Carolina, United States